CLINICAL TRIAL: NCT04143984
Title: A Phase 2 Randomized Clinical Trial to Examine the Efficacy of Carbon-Ion Radiotherapy Plus Camrelizumab As Salvage Treatment for Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: Carbon-Ion Radiotherapy Plus Camrelizumab for Locally Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Prof., Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2019-34
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Induction Chemotherapy; Heavy Ion Radiotherapy; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-C (Active Comparator): Patients will receive induction chemotherapy followed by carbon-ion radiotherapy with a dose of 63 GyE in 21 fractions (the fraction size is 3 GyE).
  Interventions: Drug: Induction chemotherapy; Radiation: Carbon-ion radiotherapy
- Arm-CC (Experimental): Patients will receive induction chemotherapy followed by carbon-ion radiotherapy and camrelizumab. In details, patients will receive carbon-ion radiotherapy with a dose of 63 GyE in 21 fractions (the fraction size is 3 GyE); in addition, patients will also receive camrelizumab of 200 mg (IV.), every 2 weeks, started with carbon-ion radiotherapy for a maximal period of 1 year.
  Interventions: Drug: Induction chemotherapy; Radiation: Carbon-ion radiotherapy; Drug: Camrelizumab

INTERVENTIONS:
Drug: Induction chemotherapy — Induction chemotherapy with the regimen of gemcitabine plus nedaplatin.
Radiation: Carbon-ion radiotherapy — Accelerated carbon-ion beam with pencil beam scanning technique.
Drug: Camrelizumab — An anti-PD-1 antibody.
  Other Names: SHR-1210
  Arms: Arm-CC

SUMMARY:
The purpose of this trial is to examine the role of camrezlizumab in addition to carbon-ion radiotherapy (CIRT) for patients with locally recurrent nasopharyngeal carcinoma. According to the plan, a total of 146 patients will be recruited and randomized into: 1) CIRT alone group (control group); 2) CIRT plus camrelizumab group (experimental group).

DETAILED DESCRIPTION:
Treatment for locally recurrent nasopharyngeal carcinoma (LR-NPC) is challenging. Carbon-ion radiotherapy appeared to be an effective treatment for this group of patients, and has substantially improved the 2-year overall survival (OS) to approximately 85%, compared to photon-based intensity-modulated radiotherapy. However, a group of the patients may still develop disease progression after CIRT, and the 2-year progression-free survival (PFS) was approximately 45%-50%. Camrelizumab, a programmed cell death 1 (PD-1) inhibitor, has been demonstrated that it is effective in the recurrent/metastatic nasopharyngeal carcinoma; however, the role of camrelizumab in concurrence with radiotherapy, especially CIRT, for LR-NPC is not clear. The purpose of this phase 2 clinical trial is to compare the efficacy of CIRT plus camrelizumab and CIRT alone in the treatment of LR-NPC. Eligible participants will be randomized (1:1) to 1) CIRT alone group (control group); 2) CIRT plus camrelizumab group (experimental group). The primary endpoint is progression-free survival. Secondary endpoints include overall survival (OS), local progression-free survival (LPFS), regional progression-free survival (RPFS), and distant metastasis-free survival (DMFS) and toxicities. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Completed a definitive course of intensity-modulated photon radiation therapy (IMRT) to a total dose of ≥ 66 Gy
* Recurrence at nasopharynx diagnosed more than 6 months after the initial course of IMRT
* Patients with neck lymphadenopathy should receive neck dissection before randomization
* With measurable lesion on contrast MR scan
* Age ≥ 18 and < 70 years of age
* ECOG score: 0-1
* Leucocyte count ≥ 4000/µL, neutrocyte count ≥ 2000/µL, platelet count ≥ 100000/µL, hemoglobin ≥ 90g/L
* Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN), alkaline phosphatase < 2.5×ULN, bilirubin ≤ ULN, serum creatinine ≤ ULN, creatinine clearance ≥ 60ml/min
* Willing to accept adequate contraception
* Ability to understand the nature of the clinical trial and sign the written informed consent

Exclusion Criteria:

* Presence of distant metastasis
* Previously received radioactive particle implantation
* Prior malignancy within 5 years before randomization, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer
* Patients who received local (such as surgery and cryotherapy) or systemic treatment, except for induction chemotherapy after diagnosis of recurrence
* With uncontrolled active infection
* With pneumonia
* With autoimmune disease
* With a known history of testing positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* Hepatitis B virus (HBV) DNA ≥ 500IU/mL for patients with positive HBV surface antigen, positive hepatitis C virus RNA for patients with positive HCV antigen
* Previously treated by immune checkpoint inhibitors
* Medical conditions requiring treatment of antibiotics and/or corticosteroid
* Treated with ≥ 5 days antibiotics one month before start of immunotherapy
* With known allergy to any of the study drugs
* Pregnant or lactating women
* Any severe intercurrent disease that may interfere with the current study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2-year
  Duration from randomization to documented disease recurrence or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 2-year
  Duration from randomization to death from any cause.
Local progression-free survival | 2-year
  Duration from randomization to documented local recurrence or death from any cause, whichever occurs first.
Regional progression-free survival | 2-year
  Duration from randomization to documented regional recurrence or death from any cause, whichever occurs first.
Distant metastasis-free survival | 2-year
  Duration from randomization to documented distant metastasis or death from any cause, whichever occurs first.
Number of participants with adverse events | 2-year
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data on participants' clinical features, treatment modalities, survivals and toxicity profile will be shared upon reasonable request. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 3 years after publication of the study.
Access Criteria: Data mentioned in the plan description and relevant supporting files will be shared with radiation oncologist who are interested in conducting pooled analysis comparing carbon-ion radiotherapy with other treatment modalities (such as other radiation technique and systemic therapy) for patients with recurrent nasopharyngeal carcinoma. The IPD will only be shared after the study protocol is reviewed and approved by the principle investigator.

REFERENCES:
- [Derived] Hu J, Huang Q, Hu W, Gao J, Yang J, Zhang H, Lu JJ, Kong L. A protocol for a randomized trial evaluating the role of carbon-ion radiation therapy plus camrelizumab for patients with locoregionally recurrent nasopharyngeal carcinoma. Cancer Med. 2024 Feb;13(3):e6742. doi: 10.1002/cam4.6742. Epub 2024 Jan 11. PMID 38205914